CLINICAL TRIAL: NCT06113211
Title: Nonopioid Pain Control Regimen After Open Reduction and Internal Fixation of Traumatic Fractures
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15315
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2024-12

CONDITIONS: Opioid Use; Fractures, Bone; Trauma
MeSH Terms: conditions — Fractures, Bone; Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Narcotic Postoperative Pain Control (Active Comparator): Standard of care control group given standard opioid pain control regimen.
  Interventions: Drug: Narcotic pain medication
- Nonnarcotic Postoperative Pain Control (Experimental): Experimental group given nonopioid pain control regimen.
  Interventions: Drug: Nonnarcotic pain medications

INTERVENTIONS:
Drug: Narcotic pain medication — Primary intervention is pain medication received postoperatively. Control group will receive the standard of care which is opioid medications. Experimental group will receive a nonopioid pain control regimen.
  Arms: Narcotic Postoperative Pain Control
Drug: Nonnarcotic pain medications — Primary intervention is pain medication received postoperatively. Control group will receive the standard of care which is opioid medications. Experimental group will receive a nonopioid pain control regimen.
  Arms: Nonnarcotic Postoperative Pain Control

SUMMARY:
An open reduction and internal fixation is a painful procedure requiring intensive postoperative pain management. Traditionally, opioid analgesia has been the gold standard for postoperative pain control. However, given the harmful side effect profile and opioid epidemic in the United States, it is advantageous to use alternate forms of analgesia. Multimodal pain control captures the effectiveness of different analgesic modalities and maximizes analgesia while minimizing side effects. The theory behind their use is that agents with different mechanisms of action work synergistically in preventing acute pain.

Objective: To measure postoperative pain control in patients in two treatment arms of ORIF of the clavicle: a treatment group given a nonopioid pain control regimen, and a standard of care control group given standard opioid pain control regimen.

Study Design: A randomized single blinded standard of care controlled clinical trial comparing pain management interventions. All adult patients scheduled for an ORIF following a traumatic fracture by fellowship trained Trauma surgeons will be eligible for inclusion. Patients will be excluded if their medical history presents known allergies or intolerance to Motrin, Lyrica, Tylenol, Zanaflex, substantial alcohol or drug abuse, and pregnancy, history of narcotics within 6 months of surgery, renal impairment, peptic ulcer disease, GI bleeding.

On the day of surgery, patients will be randomized to receive a nonopioid pain control regimen or an opioid regimen using a computer-generated sequence.

If pain is uncontrolled, patients will also be sent home with a prescription with 10 pills of 5 mg of Oxycodone for breakthrough pain. The amount of oxycodone taken will be recorded. Patients can call the resident on call, available 24-hours per day, if additional pain control is needed.

Treatment: All patients will undergo previously scheduled ORIF of the clavicle in standard fashion and be randomized to the non-narcotic pain regimen vs the narcotic pain regimen.

DETAILED DESCRIPTION:
An open reduction and internal fixation is a painful procedure requiring intensive postoperative pain management. Traditionally, opioid analgesia has been the gold standard for postoperative pain control. However, given the harmful side effect profile and opioid epidemic in the United States, it is advantageous to use alternate forms of analgesia. Multimodal pain control captures the effectiveness of different analgesic modalities and maximizes analgesia while minimizing side effects. The theory behind their use is that agents with different mechanisms of action work synergistically in preventing acute pain.

Objective: To measure postoperative pain control in patients in two treatment arms of ORIF of the clavicle: a treatment group given a nonopioid pain control regimen, and a standard of care control group given standard opioid pain control regimen.

Study Design: A randomized single blinded standard of care controlled clinical trial comparing pain management interventions. All adult patients scheduled for an ORIF following a traumatic fracture by fellowship trained Truama surgeons will be eligible for inclusion. Patients will be excluded if their medical history presents known allergies or intolerance to Motrin, Lyrica, Tylenol, Zanaflex, substantial alcohol or drug abuse, and pregnancy, history of narcotics within 6 months of surgery, renal impairment, peptic ulcer disease, GI bleeding.

On the day of surgery, patients will be randomized to receive a nonopioid pain control regimen or an opioid regimen using a computer-generated sequence.

The traditional narcotic intervention is: 60 pills of Norco 5-325 q4 hours PRN.

Patients in the nonnarcotic and narocotic intervention will be given the following pre-operative pain protocol:

Celebrex 400mg PO, Lyrica 75mg x1 dose pre-op, Tramadol 50mg x 1

Patients in the non-narcotic and narcotic intervention will be given the following intraoperative pain injection:

Epinephrine 1mg (1mL), 0.5% ropivacaine (60mL), Acetaminophen 1000mg IV, Toradol 30mg (1ml)

Postoperative day 1:

Motrin - also known as ibuprofen 800 mg every 6 hours; not to exceed 3200 mg/day

Lyrica - also known as pregabalin 75mg q12hr

Tylenol - also known as acetaminophen 1000mg PO q8hr PRN pain

Zanaflex - also know as tizanidine 4mg PO q6hr

The Postoperative pain control will be as follows:

Weeks 1 and 2:

1. Motrin - also known as Ibuprofen (for 2 weeks) 800 mg every 6 hours; not to exceed 3200 mg/day
2. Lyrica (also known as pregabalin) 75mg twice per day for 5 days then wean off as described below. Dispense: 30 tablets at discharge (75mg/tablet). Days 6-7: morning-75mg; evening- 75mg. Days 8-9: morning-75mg. Days 10: No more Lyrica
3. Tylenol (also known as acetaminophen) 1000 mg three times per day. Do not exceed a total of 4 grams of Acetaminophen per day.
4. Zanaflex (also known as tizanidine) 4 mg every 6-12 hours for 2 weeks. Weeks 2 - 4: 1. Tylenol (also known as acetaminophen) 1000 mg three times per day. Do Not exceed a total of 4 grams of Acetaminophen per day.

If pain is uncontrolled, patients will also be sent home with a prescription with 10 pills of 5 mg of Oxycodone for breakthrough pain. The amount of oxycodone taken will be recorded. Patients can call the resident on call, available 24-hours per day, if additional pain control is needed.

Treatment: All patients will undergo previously scheduled ORIF of the clavicle in standard fashion and be randomized to the non-narcotic pain regimen vs the narcotic pain regimen.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients over age eighteen and scheduled for primary open reduction internal fixation following a traumatic fracture at Henry Ford Hospital (Detroit, Michigan, United States), and Henry Ford West Bloomfield Hospital (West Bloomfield, Michigan, United States) will be eligible for inclusion in this study. All patients will be met in our abulatory orthopedic clinics. All surgeries will be performed by a fellowship trained truama surgeons.

Exclusion Criteria:

* patients with a medical history of known allergies or intolerance to allergies or intolerance to Motrin, Lyrica, Tylenol, tramadol, Zanaflex
* substantial alcohol or drug abuse
* pregnancy
* history of narcotics within 6 months of surgery
* renal impairment, peptic ulcer disease, GI bleeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Pain Score | Pain scores will be recorded daily for the first 2 weeks, and then once a week until the 6 week post operative clinic visit.
  Analog pain score 0-10. A pain score of 10 represents maximum pain and a pain score of 0 represents no pain.

SECONDARY OUTCOMES:
Patient reported function score | Preoperative visit and postoperative visits up to 1 year.
  Patient reported function questionnaire will be administered to patients during postoperative visits.

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Hospital System, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-19): https://cdn.clinicaltrials.gov/large-docs/11/NCT06113211/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-19): https://cdn.clinicaltrials.gov/large-docs/11/NCT06113211/ICF_001.pdf